CLINICAL TRIAL: NCT01539720
Title: Levonorgestrel Intrauterine System For Emergency Contraception: a Randomized Control Trial
Brief Title: Levonorgestrel Intrauterine System For Emergency Contraception
Acronym: LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of the St. Louis Region and Southwest Missouri (Other)
Collaborators: William and Flora Hewlett Foundation (Other); University of Colorado, Denver (Other); Planned Parenthood Federation of America (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201201007
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy, Unplanned; Pregnancy; Accident
Keywords: emergency contraception; Ella; Mirena IUD; post-coital contraception; Liletta IUD
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levonorgestrel Intrauterine System (Experimental): Participants randomized to the levonorgestrel IUS will undergo placement at the time of randomization. They will follow-up with a self-administered urine pregnancy test 5-6 weeks following.
  Interventions: Device: levonorgestrel IUS
- Ulipristal acetate (Active Comparator): Women in this arm will receive the oral Ulipristal acetate (Ella) regimen, which is currently the most effective method of oral emergency contraception.
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate — 30 mg tablet
  Other Names: Ella
  Arms: Ulipristal acetate
Device: levonorgestrel IUS — Levonorgestrel IUS, 52mg placed intrauterine
  Other Names: Mirena IUD; Liletta
  Arms: Levonorgestrel Intrauterine System

SUMMARY:
The purpose of this research study is to test the levonorgestrel intrauterine system as a method for emergency contraception. Emergency contraception refers to pregnancy prevention after an act of intercourse.

While the levonorgestrel intrauterine system is approved as a contraceptive method, it is considered investigational as emergency contraception, which means that it has not been approved by the U.S. Food and Drug Administration. This study will compare the device to the most common types of emergency contraception, oral Ulipristal acetate, or oral levonorgestrel. The oral levonorgestrel regimen was approved as a method of emergency contraception by the U.S. Food and Drug Administration in 1998. This method involves taking a 1.5mg pill of levonorgestrel in a single, one time dose. The Ulipristal acetate was approved as a method of emergency contraception by the U.S. Food and Drug Administration in 2010. This method involves taking a 30mg pill of Ulipristal acetate in a single, one time dose.

DETAILED DESCRIPTION:
Unintended pregnancy rates in the United States are among the highest of developed nations. These high rates can largely be attributed to incorrect or under contraception of women. One focus of decreasing unintended pregnancy and abortion rates has centered on expanding access to and use of long acting reversible contraceptive (LARC) methods which include intrauterine devices (IUDs) and subdermal implants. Emergency contraception, or post-coital contraception, offers significant reductions in the chance of pregnancy following an act of unprotected or under-protected vaginal intercourse. The most common methods of emergency contraception used in the United States are the oral levonorgestrel regimen and oral ulipristal acetate (Ella) regimen which reduce pregnancy risk by up to 89%. More effective, but rarely used, is the Cu T-380 intrauterine device (Copper IUD). The IUD has the added benefit of providing extended contraceptive use beyond the single episode of unprotected intercourse. The Cu-T380 has been associated with heavier and more crampy menses however, likely dissuading women from use. Among all IUD users, the levonorgestrel intrauterine system (LNG-IUS) has gained popularity over the Cu-T380, perhaps because it offers the potential to improve menstrual related symptoms. There is no data however on the efficacy of the LNG-IUS as a form of emergency contraception. The purpose of this study is to evaluate the efficacy of the LNG-IUS as a method of emergency contraception. Participants will be randomized to receive either the most common method, oral emergency contraception, or the LNG-IUS. Participants will then be evaluated 5-6 weeks following method allocation for pregnancy. Lastly, participants will be asked to complete a telephone surveys at 6 and 12 months following method allocation assessing their use of a consistent contraceptive method, their satisfaction with their contraceptive method, any use of emergency contraception since their enrollment in the study, and lastly any unintended pregnancies experienced since enrollment in the study. If we could show that the LNG-IUS is as effective as the most commonly prescribed method of emergency contraception, we would be introducing another opportunity for LARC initiation and subsequently impacting unintended pregnancy and abortion rates.

ELIGIBILITY:
Inclusion Criteria:

* Women age 14-45
* Under-protected intercourse within the last five days (120 hours)
* Willingness to accept either intervention: intrauterine contraception or oral emergency contraception (EC)
* Ability and willingness to follow-up for in clinic urine pregnancy test (UPT)
* Ability and willingness to be contacted by phone for 6 and 12 month follow-up

Exclusion Criteria:

* Positive pregnancy test
* Non-English speaking
* Contraindication to intrauterine contraception or oral EC
* Inability or unwillingness to comply with follow-up

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 274 (Actual)
Dates: Start 2012-12; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McNicholas, DO, MCSI, Principal Investigator — Planned Parenthood of the St. Louis Region and Southwest Missouri
Locations (3):
- United States (3):
  - Atlanta Women's Center, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University School of Medicine in St. Louis, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levonorgestrel Intrauterine System | Ulipristal Acetate
Started | 198 | 76
5 WEEKS | 183 | 73
6 MONTHS | 169 | 66
Completed | 169 | 66
Not Completed | 29 | 10
Not completed — Screen Fail | 15 | 3
Not completed — Lost to Follow-up | 14 | 7

BASELINE CHARACTERISTICS:
Population: We randomized 274 participants in the study, of which 256 completed five-week follow-up, and 235 (85.8%) had complete six month follow-up data. The baseline demographics are based on the 256 participants who were available for analysis after completion of the 5 week follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Levonorgestrel Intrauterine System | Ulipristal Acetate | Total
Number analyzed (Participants) | 183 | 73 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 73 | 256
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (6.1) | 27.1 (6.5) | 27.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 73 | 256
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 5 | 20
  Not Hispanic or Latino | 168 | 68 | 236
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 66 | 40 | 106
  White | 93 | 26 | 119
  Other | 23 | 7 | 30
  Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 183 | 73 | 256

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pregnancy Following Emergency Contraception
Description: Observed pregnancies at 5 weeks and at 6 months in the LNG-IUD group will be compared to those in the oral UPA group.
Time Frame: 5 weeks post-randomization
Population: total eligible for analysis after 5-6 weeks post randomization = 256; total eligible for analysis after 6 months post randomization = 235
Measure: Count of Participants; unit: Participants
Arm/Group | Levonorgestrel Intrauterine System | Ulipristal Acetate
Number analyzed (Participants) | 183 | 73
Participants
  Pregnancy at 5 weeks post randomization. | 0 | 0
  Pregnancy at 6 months post randomization.: number analyzed (Participants) | 169 | 66
  Pregnancy at 6 months post randomization. | 0 | 6

2. Secondary Outcome: Number of Participants Using Any LARC Method at 6 Months Post Randomization
Description: The number of participants who reported using any type of long acting reversible contraception (LARC) use at 6 months following method allocation will be evaluated, whether or not it was their allocated LNG-IUS.
Time Frame: 6 months post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Levonorgestrel Intrauterine System | Ulipristal Acetate
Number analyzed (Participants) | 169 | 66
Participants | 95 | 13

3. Secondary Outcome: Number of Participants Reporting Continuation and Satisfaction With Their Study Allocated LNG-IUS
Description: Continuation and satisfaction among participants in the LNG-IUS arm who reported still using their LNG-IUS at 6 month post randomization.
Time Frame: 6 months post randomization
Population: 169 = total eligible for analysis from randomized LNG-IUS arm; at 6 months post randomization, 92 of 169 were still using LNG-IUS, so only 92 eligible to analyze satisfaction with LNG-IUS at 6 months post randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Levonorgestrel Intrauterine System
Number analyzed (Participants) | 169
Participants
  Continuation of LNG-IUS at 6 months | 92
  Satisfaction with LNG-IUS at 6 months: number analyzed (Participants) | 92
  Satisfaction with LNG-IUS at 6 months | 82

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Levonorgestrel Intrauterine System | Ulipristal Acetate
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/73
Other Adverse Events (participants affected / at risk) | 0/183 | 0/73

LIMITATIONS AND CAVEATS:
Group size limits the precision of our estimate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT01539720/Prot_SAP_000.pdf